CLINICAL TRIAL: NCT02189915
Title: Open-Label Creatine Monohydrate Supplementation in Depressed Female Methamphetamine Users
Brief Title: Open-Label Creatine Study for Female Meth Users
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Received funding for the next phase of the study
Sponsor: Perry Renshaw (Other)
Responsible Party: Sponsor-Investigator, Perry Renshaw, Professor of Psychiatry, University of Utah
Organization: University of Utah (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 53737
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Results first posted 2016-05-20 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-04

CONDITIONS: Depression; Dual Diagnosis; Substance Use
MeSH Terms: conditions — Depression; Substance-Related Disorders | interventions — Creatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Creatine monohydrate (Experimental)
  Interventions: Drug: Creatine monohydrate

INTERVENTIONS:
Drug: Creatine monohydrate

SUMMARY:
Study Purposes and Objectives:

The objectives should be stated in such a way that the reader can determine the appropriateness of the study design. If appropriate, state the specific hypotheses being tested and/or study aims. Use lay language.

Methamphetamine use is of great concern in the state of Utah because it's the primary drug of threat in the state, and is the primary drug of choice among females between the ages of 18 and 24. The primary hypothesis of the study is that eight weeks of oral creatine supplementation will result in improvements in depression rating scores in female MA users. Secondary hypotheses include the following: 1) creatine supplementation will result in a decrease in the number of positive MA screens; 2) NAA and Cr concentrations will increase after eight weeks of oral creatine supplementation; and 3) PCr/β-NTP levels in the frontal lobe using 31P MRS will increase after eight weeks of creatine monohydrate oral supplementation.

ELIGIBILITY:
Inclusion Criteria:

1. Must be female
2. Must be between the ages of 13 and 55 years
3. Methamphetamine must be primary drug of choice
4. Must have used methamphetamine within the last 6 months
5. For participants > 18 years of age, must have a Hamilton Depression Rating Scale (HDRS or HAM-D) score of > 17
6. For participants < 18 years of age, must have a Children Depression Rating Scale (CDRS) score of > 40
7. Must be able to give informed consent

Exclusion Criteria:

1. Significant current or past medical conditions, such as cardiovascular, renal or endocrine disorders
2. DSM-IV diagnosis of bipolar disorder, schizophrenia, or schizoaffective disorder
3. Known pregnancy or positive urine HCG test
4. Current serious homicidal or suicidal risk
5. Young Mania Rating Scale (YMRS) score > 7
6. Inability to comply with the protocol
7. Contraindication to an MR scan
8. Positive HIV test
9. Known sensitivity to creatine monohydrate

Inclusion criteria for healthy comparison group:

1. Must be female
2. Must be between the ages of 13 and 55 years
3. Must be able to give informed consent

Exclusion criteria for healthy comparison group:

1. Significant current medical illness
2. DSM-IV disorder identified by the SCID (to include bipolar I, bipolar II, bipolar NOS, major depressive disorder, dysthymia disorder, depressive disorder NOS, primary psychotic symptoms, substance use disorders, and anxiety disorders)
3. Known pregnancy or positive urine HCG test
4. Contraindication to an MR scan
5. Inability to comply with the protocol
6. Positive urine drug screen (unless it is positive for a low dose prescription opiate that is taken as prescribed)

Ages: 13 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2012-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perry Renshaw, MD, PhD, MBA, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Creatine Monohydrate Treatment: This study is an open label study, where all participants received Creatine monohydrate.
Period: Overall Study
Arm/Group | Creatine Monohydrate Treatment
Started | 14
Completed | 11
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Creatine Monohydrate: Creatine monohydrate
Arm/Group | Creatine Monohydrate
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Depression Rating Scores
Description: Hamilton Depression Rating Scale scores is used to assess the level of depression. The Hamilton Depression Rating Scale ranges from 0 to 50. A score of 0-7 is considered to be normal. A score of 8-13 indicates mild depression. A score of 14-18 indicates moderate depression. Scores higher than 19 indicate severe depression.
Time Frame: 8-week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Creatine Monohydrate Treatment
Number analyzed (Participants) | 11
units on a scale
  Baseline | 16.86 (3.40)
  After 8 weeks of treatment | 7.36 (4.59)

2. Secondary Outcome: Phosphocreatine Levels Measured by Magnetic Resonance Spectroscopy
Description: Phosphocreatine (PCr) was measured pre- and post-creatine treatment to assess changes in neurochemistry. Creatine treatment may increase brain intracellular PCr, and brain energy metabolism has been suggested to play a role in the pathophysiology of depression. Increased levels of PCr suggest reduced depressive symptoms. PCr levels are calculated using a ratio and remains unitless.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Phosphocreatine levels (unitless)
Arm/Group | Creatine Monohydrate Treatment
Number analyzed (Participants) | 10
Phosphocreatine levels (unitless)
  Baseline | 0.223 (0.013)
  Post-treatment | 0.233 (0.009)

ADVERSE EVENTS:
Arm/Group | Creatine Monohydrate Treatment
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 14/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Creatine Monohydrate Treatment (N=14)
Flu like symptoms (General disorders) | 13
Indigestion, Nausea (Gastrointestinal disorders) | 6
Numbness, tingling (Nervous system disorders) | 1
Swelling in hands (General disorders) | 4
Blurry vision (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No